CLINICAL TRIAL: NCT05342519
Title: Daily Topical Rapamycin Therapy for the Treatment of Vitiligo
Brief Title: Daily Topical Rapamycin for Vitiligo
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: American Skin Association (Other)
Responsible Party: Principal Investigator, Chelsea Shope, Medical/Dental Resident, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115924
Record Dates: First submitted 2022-04-19; First posted 2022-04-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Vitiligo
Keywords: Dermatology; Pediatrics; Rapamycin
MeSH Terms: conditions — Vitiligo | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: During a clinical care visit, if a patient is eligible and agrees to participate, one lesion occupying less than 2% body surface area (BSA) will be identified for treatment with either 0.1% or 0.001% topical rapamycin cream to be applied daily for 6 months. Ten patients will be randomized to each treatment arm, however, if it is clear that one treatment arm is less effective, that treatment arm will be dropped, and study participants will be reallocated to the more effective treatment arm. A second, symmetric lesion about the same size and evolution time occupying less than 2% BSA will be identified for treatment with topical placebo cream to be applied daily for 6 months. The second lesion must be at the corresponding anatomic location on the other half of the body, i.e., if topical rapamycin is applied to the left arm, topical placebo will be applied to the right arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The pharmacy will distribute medications in unlabeled, 60-gram tubes following patient enrollment. Tubes will be marked as "Left" and "Right." The association between tube label and treatment type will only be known to pharmacy staff. The pharmacy staff will allocate 10 patients to receive 0.001% rapamycin and 10 patients to receive 0.1% rapamycin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Topical rapamycin 0.001% (Experimental): Patients randomized to this arm of the study will apply 2 finger tip units (FTU) or 0.5 cc topical rapamycin 0.001% cream daily for 6 months
  Interventions: Drug: Rapamycin
- Topical rapamycin 0.1% (Active Comparator): Patients randomized to this arm of the study will apply 2 FTU (0.5 cc) topical rapamycin 0.1% cream daily for 6 months
  Interventions: Drug: Rapamycin
- Placebo (Placebo Comparator): All patients will apply 2 FTU (0.5 cc) topical placebo cream daily for 6 months to the corresponding anatomic location on the opposite side of the body where the experimental drug is not being applied
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapamycin — While rapamycin is not approved for the treatment of vitiligo, it has been found to be efficacious in stopping disease progression in animal models. Another recent study in humans showed that doses of 0.5cc daily of 0.001% of the topical formulation are able to achieve improvement in hypopigmented lesions of the skin at both the clinical and histological level. At this dose, improvement in cell function was observed regarding maintenance of proliferative potential and prevention of senescence, with avoidance of total inhibition of cell growth as has been seen at higher potencies used for immunosuppression.
  Other Names: Sirolimus, rapamune
  Arms: Topical rapamycin 0.001%
Drug: Rapamycin — Rapamycin is an immunosuppressant that works by inhibiting the mammalian target of rapamycin (mTOR) leading to inhibition of the cell cycle and antibody production. It has also been shown to promote expansion of Treg populations. Although studies evaluating alternative dosing for vitiligo are limited, topical rapamycin has previously been used to treat angiofibromas related to Tuberous Sclerosis, vascular malformations such as port-wine stains, and inflammatory lesions such as plaque psoriasis. In a 2019 meta-analysis, 38 out of 40 reports included used topical formulations of 1% or lower potency rapamycin; the majority of publications were focused on the treatment of Tuberous Sclerosis, where the median concentration of mTOR inhibition was 0.1% dosed twice daily.
  Other Names: Sirolimus, rapamune
  Arms: Topical rapamycin 0.1%
Drug: Placebo — All patients will be assigned to received topical placebo cream to the lesion not being treated with the active study drug.
  Arms: Placebo

SUMMARY:
In current Dermatology practice, options for vitiligo remain limited. The purpose of this study is to determine if once daily dosed topical rapamycin is effective for the treatment of patients with vitiligo. Participants will apply either 0.1% topical rapamycin or 0.001% topical rapamycin for six months to a lesion on one side of the body, and topical placebo to a corresponding lesion on the opposite side of the body. The study also aims to evaluate patient satisfaction and identify any adverse effects on these dosing regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients 13 years of age and older
* Patients with nonsegmental vitiligo

Exclusion Criteria:

* Patients with segmental or mucosal vitiligo
* Patients with contraindication to use of rapamycin
* Patients with history of transplant
* Patients with a history of natural immunodeficiency
* Patients with a history of artificially induced immunodeficiency
* Patients with a history of a serious or life-threatening infection
* Patients taking CYP3A4 inhibiting medications
* Patients taking strong CYP3A4 inducers
* Patients undergoing current treatment for vitiligo
* Women that are or may become pregnant

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of lesions with no response | 6 months
  Absence of change in appearance of targeted lesion. Vitiligo is a depigmenting disease and treatment responses are graded by percentage of repigmentation on a 5-point scale
Number of lesions with partial response | 6 months
  There is change in the size of dyspigmentation as compared to its appearance and symptoms at the initial visit, but the lesion remains grossly visible. Vitiligo is a depigmenting disease and treatment responses are graded by percentage of repigmentation on a 5-point scale. Changes in the characteristics of the targeted lesions will be evaluated by a dermatologist and documented via photographs at follow-up visits at 2, 4, and 6-months, with the final outcome measured at the 6-month visit.
Numbers of lesions with complete response | 6 months
  Targeted lesion is no longer grossly visible.

SECONDARY OUTCOMES:
Average score of Dermatology Quality of Life questionnaire (or Teenager Quality of Life Index) | 6 months
  The Dermatology Life Quality Index (DLQI) is designed to measure the health-related quality of life of adult (or teenage) patients suffering from a skin disease. Both physical and psychological symptoms are ranked on a 4-point scale from "not at all" to "very much" to provide a cumulative patient score.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Aleisa, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No